CLINICAL TRIAL: NCT00154622
Title: National Taiwan University Hospital
Brief Title: Management and Outcome of Work-Related Musculoskeletal Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 9261701040; DOH94-HP-1405
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Neck Injury; Back Injury; Arms Injury; Cumulative Disorder
Keywords: musculoskeletal disorder, work hardening, return to work
MeSH Terms: conditions — Neck Injuries; Back Injuries; Musculoskeletal Diseases

ARMS (1):
- pain/ disability survey (No Intervention)
  Interventions: Behavioral: work hardening program

INTERVENTIONS:
Behavioral: work hardening program

SUMMARY:
Work-related musculoskeletal disorders(MSD)are very common，which account for most of the occupational compensation in U.S.A。According to the epidemiological surveys，injured sites are frequent at low back，neck and shoulder and upper extremity。Although the MSD will not threaten the lives，they result in discomfort，some cost much and decrease the productivity。There was little study in our country to reveal the risk factors of medical utilization and disabling of MSD。Therefore，we do not have well-established strategy of the assessment and treatment for the workers who can not return to work。The purposes of this study are：1、To have sequential surveys to find the prevalence，incidence and possible risk factors of work-related MSD of employees in different industries and their medical utilization and disabled conditions。2、To find the victims of work-related MSD from clinics，assess their disablement and if they return to work and to find the factors those prevent them return to work。3、To develop individualized work hardening programs for the victims who can not return to wok after treatment。The program will be established according to their injuries and their work characteristics。

DETAILED DESCRIPTION:
Work-related musculoskeletal disorders(MSD)are very common，which account for most of the occupational compensation in U.S.A。According to the epidemiological surveys，injured sites are frequent at low back，neck and shoulder and upper extremity。Although the MSD will not threaten the lives，they result in discomfort，some cost much and decrease the productivity。There was little study in our country to reveal the risk factors of medical utilization and disabling of MSD。Therefore，we do not have well-established strategy of the assessment and treatment for the workers who can not return to work。The purposes of this study are：1、To have sequential surveys to find the prevalence，incidence and possible risk factors of work-related MSD of employees in different industries and their medical utilization and disabled conditions。2、To find the victims of work-related MSD from clinics，assess their disablement and if they return to work and to find the factors those prevent them return to work。3、To develop individualized work hardening programs for the victims who can not return to wok after treatment。The program will be established according to their injuries and their work characteristics。In the first year，questionnaire will be used to find the prevalence of work-related MSD of employees in different industries with various work types。The demographic factors and the exposure factors will also be collected to find the risk factors。One month and 6 months after the first surveillance，the 2nd and 3rd surveillances will be executed to find the new incidence and their medical utilization and loss of work time。In the second year，the injured workers（in low back，neck and shoulder and upper extremity）from outpatient departments will be followed and assessed。They will be followed for 3 months to reveal their medical need，their recovery and if they return to work after treatment。According to all the data，we can find the ratios of loss of work time in different types of injuries and the risk factors causing unable to return to work。In the second half of this year，the authors will begin to establish the individualized work hardening programs and to finish the prevention and training booklets。In the third year，we will find the workers who can not return to wok after 3-month treatment in the clinics。After the assessment of their severity and residual working ability，the workers will be randomized into training or control groups。There will be 15 workers in each group in 3 kinds of injuries（low back，neck and shoulder and upper extremity），totally 90 workers will be recruited。After 3-month work hardening training program，re-assessment will be done and their return-to-work rate will be followed 3 and 6 months later。

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 65 years have a job

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2004-01; Primary Completion 2006-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
functional capability evaluation | referral to and duration of PT at the the first day
pain evaluation | referral to and duration of PT at the the first day

CONTACTS AND LOCATIONS:
Overall Officials: J Y Tsauo, PhD, Study Director — Grad School of PT, College of Medicine, NTU
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan